CLINICAL TRIAL: NCT00065403
Title: Acupuncture for Irritable Bowel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT001414 (NIH); KaptchukTJ
Record Dates: First submitted 2003-07-22; First posted 2003-07-23 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Acupuncture
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Acupuncture Therapy

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
Little is known about acupuncture's efficacy for Irritable Bowel Syndrome (IBS). This trial uses a manualized acupuncture treatment format that closely follows clinical practice and allows flexibility in designing individualized treatments. In addition, a second parallel qualitative study will follow a subgroup of patients throughout the trial to explore the relationships between patients' interpretations and understandings (what anthropologists call "meaning") of irritable bowel and their response to treatment. Cortisol levels (an important stress hormone) will also be assessed.

This will be a 3-arm trial: Active acupuncture, placebo acupuncture, and wait list.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of Irritable Bowel Syndrome based on Rome II criteria, including at least 12 weeks of abdominal discomfort or pain in the last 12 months with at least 2 of the following features:

* Relief with defecation
* Onset associated with a change in stool frequency
* Onset associated with a change in form/appearance of stool

Exclusion criteria:

* History of severe or intractable IBS, defined as continuous, unremitting and several abdominal pain greater than 12 hours/day
* Previous acupuncture treatment
* Concurrent diagnosis of any bowel disturbance that would interfere with the assessment or safety of the study
* History of laxative abuse
* Previous abdominal surgery (uncomplicated appendectomy, hysterectomy or cholecystectomy at least 6 months prior to entry acceptable)
* History of metabolic or inflammatory disease that may affect bowel motility, eg.g., inflammatory bowel disease, diabetes mellitus, sarcoidosis
* Other significant illness as determined by Investigator
* History of drug or alcohol abuse w/in 2 years;
* Insufficient knowledge of English to complete self-assessments to participate in study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2004-02; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Ted Kaptchuk, OMD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493